CLINICAL TRIAL: NCT04805853
Title: Myocardial Pathological Changes in Patients of Type 2 Diabetes With or Without PCOS Using Cardiac Magnetic Resonance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2020-198
Record Dates: First submitted 2021-03-02; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Type2 Diabetes; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Whole blood,fasting serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- type 2 diabetes without polycystic ovary syndrome: The treatment of type 2 diabetes is based on the Chinese Medical Association Diabetes Branch '2017 China Type 2 Diabetes Prevention Guidelines' for lifestyle adjustment and diabetes drug treatment.The research physician decides the diabetes treatment measures of the research object; the blood sugar control goal is that glycosylated hemoglobin is less than 7%.
- polycystic ovary syndrome without type 2 diabetes: The treatment of polycystic ovary syndrome is based on the '2018 Polycystic Ovary Syndrome Chinese Diagnosis and Treatment Guidelines' by the Endocrinology Group of the Obstetrics and Gynecology Branch of the Chinese Medical Association and the Guide Expert Group '2018 Polycystic Ovary Syndrome Expert consensus on diagnosis and treatment of endocrinology' for lifestyle and drug treatment.
- polycystic ovary syndrome with type 2 diabetes: Treatment is as above.

SUMMARY:
The study is prepared to use CMR technology for early screening of myocardial lesions in 561 age-matched women with type 2 diabetes without PCOS, with PCOS without type 2 diabetes and with type 2 diabetes combined with PCOS, compare the differences between the two groups of cardiomyocyte injury changes, and treat and follow-up with type 2 diabetes and PCOS in accordance with the current standard treatment guidelines for type 2 diabetes and PCOS, after 3 years of follow-up we will analyse the changes in cardiomyopathy, cardiac serological indicators, and heart function indicators,which can provide theoretical basis for early clinical intervention in the future.

DETAILED DESCRIPTION:
So far, due to the lack of more sensitive noninvasive detection methods and indicators that suggest early cardiomyopathy, it is not clear whether type 2 diabetes combined with PCOS will lead to earlier and more progressive changes in cardiomyopathy, and whether there is a difference with type 2 diabetes alone and early cardiomyopathy in patients with simple PCOS.Compared with women with type 2 diabetes who did not combine polycystic Ovary Syndrome(PCOS) or PCOS did not combine with type 2 diabetes, patients with type 2 diabetes who combined PCOS had the characteristics of lower age of onset, longer exposure to high risk factors of CVD, and higher risk of cardiovascular disease on the basis of the dual pathophysiology of insulin resistance and hyperandrogenism.The purpose of this study is to find early cardiovascular disease of women with type 2 diabetes and PCOS and conduct early clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-40 years old;
2. Overweight and obese women with/without type 2 diabetes without PCOS, PCOS without type 2 diabetes, and type 2 diabetes with PCOS;
3. HbA1C 7-9% of patients with type 2 diabetes;
4. Increased risk of cardiovascular disease (with any one of the following risk factors: hypertension, dyslipidemia, hyperuricemia, obesity, smoking);
5. The diagnosis of PCOS is based on the 2003 Rotterdam criteria, the diagnosis of overweight/obesity is based on the WHO-WPR criteria, and the diagnosis criteria of type 2 diabetes is based on the 1998 WHO diagnosis criteria;
6. Willing to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Severe liver and kidney dysfunction (ALT is greater than 2.5 times the upper limit of normal, or Cr>132umol/l, or eGFR <60 mL/min/1.73m2), psychosis, accompanied by severe infection, severe anemia, neutropenia disease;
2. Congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, atrial fibrillation, viral myocarditis, infectious myocarditis, hyperthyroid heart disease, cardiac amyloidosis and other myocardial damage diseases, NYHA heart function classification ≥ Grade III, or the subject has had a clinical cardiovascular event in the past 3 months;
3. Symptomatic heart failure in the past 6 months, or left ventricular ejection fraction <35%;
4. Self-reported or medical records are type 1 diabetes, single-gene mutation diabetes, diabetes caused by pancreatic injury, or other secondary diabetes (such as diabetes caused by Cushing syndrome, abnormal thyroid function, or acromegaly) ；
5. Pregnancy;
6. Participated in clinical trials of other drugs within 3 months;
7. In the past 5 years, there have been treated or untreated organ system tumors (except local skin basal cell carcinoma), regardless of whether there is evidence of local recurrence or metastasis;
8. A history of psychoactive substance abuse, including alcohol and a history of alcohol-related illnesses in the past 2 years;
9. The subject is allergic to the contrast agent (gadopentetate meglumine injection);
10. The subject has claustrophobia;
11. The subject contains metal implants that are not suitable for cardiac magnetic resonance examination;
12. Any conditions judged by the investigator that affect enrollment.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Overweight/obese women with type 2 diabetes without PCOS, PCOS without type 2 diabetes, and type 2 diabetes with PCOS were expected enrolled in our study.
Sampling Method: Probability Sample
Enrollment: 561 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
the change level of cardiac extracellular volume (ECV) | 3 years
  Compared with baseline, the change level of cardiac extracellular volume (ECV) in patients with type 2 diabetes without PCOS, PCOS without type 2 diabetes, and type 2 diabetes with PCOS

SECONDARY OUTCOMES:
change in the level of troponin I (TNI) | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the serum index related to myocardial injury such as change of TNI in ng/ml.
change in the level of creatine kinase isoenzymes (CK-MB) | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the serum index related to myocardial injury such as change of CK-MB in IU/L.
change in the level of Brain Natriuretic Peptide (BNP) | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the serum index related to myocardial injury such as change of BNP in pg/ml.
change in the level of atrialnatriureticpeptide (ANP) | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the serum index related to myocardial injury such as change of ANP in pg/ml.
change in the level of left ventricular ejection fraction (LVEF) | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the cardiac functions change such as: left ventricular ejection fraction (LVEF) in %.
change in the level of left ventricular end diastolic pressure (LVEDP) | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the cardiac functions change such as: left ventricular end diastolic pressure (LVEDP) in kPa/mmHg.
change in the level of output per minute (CO) in L/min | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the cardiac functions change such as: output per minute (CO) in L/min.
change in the level of left ventricular diameter reduction rate (FS) | 3 years
  Compared with the baseline in three groups and T2DM with different phenotype of PCOS, the cardiac functions change such as: left ventricular diameter reduction rate (FS) in %.
Changes in score of Minnesota heart failure quality of life scale(LiHFe) | 3 years
  Compared with the baseline in three groups, the changes of Minnesota heart failure quality of life scale(LiHFe) in score, higher scores mean a worse outcome. (Scores ranging from 0 to 105)
Changes in score of short form 12 questionnaire(SF-12) | 3 years
  Compared with the baseline in three groups, the changes of SF-12 in score, higher scores mean a better outcome. (Scores ranging from 0 to 65)
Changes in score of Generalized Anxiety Disorder-7(GAD-7) | 3 years
  Compared with the baseline in three groups, the changes of GAD-7 in score, higher scores mean a worse outcome. (Scores ranging from 0 to 21)
Changes in score of Patient Health Questionnaire-9(PHQ-9) | 3 years
  Compared with the baseline in three groups, the changes of PHQ-9 in score, higher scores mean a worse outcome. (Scores ranging from 0 to 27)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, Dr., Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Department of Endocrinology and Metabolism, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodarzi MO, Dumesic DA, Chazenbalk G, Azziz R. Polycystic ovary syndrome: etiology, pathogenesis and diagnosis. Nat Rev Endocrinol. 2011 Apr;7(4):219-31. doi: 10.1038/nrendo.2010.217. Epub 2011 Jan 25. PMID 21263450
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Mahalingaiah S, Diamanti-Kandarakis E. Targets to treat metabolic syndrome in polycystic ovary syndrome. Expert Opin Ther Targets. 2015;19(11):1561-74. doi: 10.1517/14728222.2015.1101067. Epub 2015 Oct 21. PMID 26488852
- [Background] Lim SS, Davies MJ, Norman RJ, Moran LJ. Overweight, obesity and central obesity in women with polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2012 Nov-Dec;18(6):618-37. doi: 10.1093/humupd/dms030. Epub 2012 Jul 4. PMID 22767467
- [Background] Baldani DP, Skrgatic L, Goldstajn MS, Vrcic H, Canic T, Strelec M. Clinical, hormonal and metabolic characteristics of polycystic ovary syndrome among obese and nonobese women in the Croatian population. Coll Antropol. 2013 Jun;37(2):465-70. PMID 23940991